CLINICAL TRIAL: NCT00752609
Title: A Phase 2 Study of the Safety and Efficacy of Hematide Injection for the Maintenance Treatment of Anemia in Subjects With Chronic Renal Failure Who Are on Hemodialysis or Do Not Require Dialysis and Previously Treated With Darbepoetin Alfa
Brief Title: Safety and Efficacy of Peginesatide Injection for the Maintenance of Anemia in Chronic Renal Failure Participants Who Are on Hemodialysis or Do Not Require Dialysis and Previously Treated With Darbepoetin Alfa.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFX01_202; 2008-003459-64 (EudraCT Number); U1111-1114-1500 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-06

CONDITIONS: Anemia
Keywords: Anemia; Drug Therapy; Hemodialysis; Kidney Failure
MeSH Terms: conditions — Anemia; Renal Insufficiency | interventions — peginesatide; hematide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peginesatide (Experimental)
  Interventions: Drug: Peginesatide

INTERVENTIONS:
Drug: Peginesatide — Peginesatide 0.04 to 0.16 mg/kg, subcutaneous or intravenous injection, once every 4 weeks for up to 24 weeks. Initial dose based on patient's previous total weekly darbepoetin alfa dose, and thereafter could be adjusted to maintain hemoglobin values in the target range of 10 to 12 g/dL and ±1.5 g/dL from Baseline.
  Other Names: Hematide; AF37702; Omontys

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Peginesatide Injection for the maintenance of anemia in patients with chronic renal failure who are on hemodialysis or do not require dialysis and who were previously treated with Darbepoetin Alfa.

DETAILED DESCRIPTION:
Anemia, resulting primarily from insufficient production of erythropoietin to support erythropoiesis, is a common consequence of chronic renal failure. Both North America and Europe have established clinical practice guidelines for the treatment and hemoglobin targets in chronic renal failure/chronic kidney disease patients. These guidelines recommend the use of erythropoiesis-stimulating agents (ESAs). The benefits of ESA therapy include reduced fatigue, improved quality of life, decreased cardiovascular mortality risk and improved cardiovascular function. An increased risk of death and serious cardiovascular and thromboembolic events, including myocardial infarction, stroke, congestive heart failure, and hemodialysis graft occlusion have been observed in controlled clinical trials of ESAs when administered to target hemoglobin levels of ≥13.5 g/dL. The vast majority of patients receiving hemodialysis receive ESA therapy to treat their anemia and most patients begin ESA therapy prior to any requirement for dialysis.

Anemia of chronic renal failure is due to several factors, primarily the inability of the diseased kidneys to produce adequate amounts of endogenous erythropoietin. Ancillary factors also include the shortened lifespan of red blood cells, iron and other nutritional deficiencies, infection, and inflammation. The prevalence of anemia increases with progressive deterioration of renal function, and affects more than 90% of patients with chronic renal failure Stage 5 (End Stage Renal Disease). Anemia is associated with increased mortality, increased likelihood of hospitalization, reduced cognitive function and exercise capacity, increased left ventricular hypertrophy and heart failure. Treatment of anemia reduces morbidity and mortality risks and may improve quality of life.

Erythropoiesis stimulating agents have been established as a treatment for anemia in chronic renal failure participants, and have improved the management of anemia over alternatives such as transfusion. Peginesatide (hematide) is a parenteral formulation being developed for the correction of anemia in patients with chronic renal failure, and binds to and activates the human erythropoietin receptor and stimulates erythropoiesis in human red cell precursors in a manner similar to other known erythropoiesis-stimulating agents.

Participants in this study received variable doses of peginesatide injection once every four weeks. Total commitment time for this study was about 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was a man or woman 18 to 90 years of age, inclusive.
2. The patient had CKD and met 1 of the following criteria:

   1. Had been on dialysis for ≥6 months prior to enrollment, or
   2. Had not yet begun dialysis (hemodialysis or peritoneal dialysis) and was not anticipated to require initiation of dialysis during participation in the study.
3. The patient was on stable darbepoetin alfa maintenance therapy (either SC or IV) continuously for a minimum of 8 weeks prior to enrollment.
4. The patient had 4 consecutive Hb values with a mean ≥10.0 and ≤12.0 g/dL during screening period, with the difference between the mean of the first 2 consecutive Hb values and the mean of the last 2 consecutive values being ≤1.0 g/dL.

Exclusion Criteria:

1. The patient had known bleeding or coagulation disorder.
2. The patient had known hematologic disease or cause of anemia other than renal disease (i.e., pure red cell aplasia, homozygous sickle-cell disease, thalassemia, multiplemyeloma, hemolytic anemia, and myelodysplastic syndrome).
3. The patient had received a recent course of intensive iron replacement (i.e., more than 500 mg IV in the 28 days prior to enrollment).
4. The patient had advanced chronic CKD defined by New York Heart Association Class III or IV.
5. The patient had a known history of seizure disorder or received antiepileptic medication for a seizure disorder within 6 months prior to enrollment.
6. The patient had a scheduled kidney transplant. Patients currently on a transplant waiting list were not excluded, unless there was an identified donor.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (10):
- United States (10):
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - Middlebury, Connecticut
  - Lauderdale Lakes, Florida
  - Shreveport, Louisiana
  - Dearborn, Michigan
  - Columbus, Mississippi
  - Mineola, New York
  - Arlington, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 18 investigative sites in the United Kingdom, Italy, Australia, and the United States from 22 September 2008 to 24 December 2009.
Pre-assignment Details: Participants with a diagnosis of chronic renal failure (on hemodialysis or not on dialysis) and receiving stable Darbepoetin alfa maintenance therapy were enrolled into one treatment group (peginesatide injection).
Groups:
- Peginesatide - On Dialysis: Participants on dialysis received peginesatide 0.04 to 0.16 mg/kg, subcutaneous or intravenous injection, once every 4 weeks for up to 24 weeks. Initial dose based on patient's previous total weekly darbepoetin alfa dose, and thereafter could be adjusted to maintain hemoglobin values in the target range of 10 to 12 g/dL and ±1.5 g/dL from Baseline.
- Peginesatide - Not on Dialysis: Participants not on dialysis received peginesatide 0.04 to 0.16 mg/kg, subcutaneous or intravenous injection, once every 4 weeks for up to 24 weeks. Initial dose based on patient's previous total weekly darbepoetin alfa dose, and thereafter could be adjusted to maintain hemoglobin values in the target range of 10 to 12 g/dL and ±1.5 g/dL from Baseline.
Period: Overall Study
Arm/Group | Peginesatide - On Dialysis | Peginesatide - Not on Dialysis
Started | 53 | 49
Full Analysis Set | 52 (One patient withdrew consent before receiving any study medication.) | 49
Completed | 44 | 47
Not Completed | 9 | 2
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 0
Not completed — Met exclusion criteria | 1 | 0
Not completed — Received Aranesp in error | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginesatide - On Dialysis | Peginesatide - Not on Dialysis | Total
Number analyzed (Participants) | 52 | 49 | 101
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline characteristics are reported for the Full Analysis Set.
  years | 66.4 (12.60) | 68.6 (12.07) | 67.5 (12.33)
Age, Customized [Number; unit: participants]
  < 65 years | 22 | 18 | 40
  ≥65 - <75 years | 13 | 13 | 26
  ≥ 75 | 17 | 18 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 33 | 50
  Male | 35 | 16 | 51

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Between Baseline and the Evaluation Period
Description: Mean change in Hemoglobin between Baseline (the mean of the 4 most recent hemoglobin values prior to enrollment and the hemoglobin on the day of enrollment) and the Evaluation Period (mean hemoglobin from Weeks 19 to 24).
Time Frame: Baseline and Week 19 to Week 24.
Population: The Full Analysis Set including all patients who received at least 1 dose of study drug where data was available (indicated by N).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Peginesatide - On Dialysis | Peginesatide - Not on Dialysis
Number analyzed (Participants) | 52 | 49
g/dL
  Baseline [N=52, 49] | 11.22 (0.514) | 11.11 (0.447)
  Evaluation Period [N=45, 47] | 10.78 (0.845) | 11.64 (0.673)
  Change from Baseline [N=45, 47] | -0.42 (0.761) | 0.49 (0.769)
Statistical Analysis 1: Comparison: Peginesatide - On Dialysis; Test type: Superiority or Other; Mean change from baseline = -0.42, 95% CI 2-sided [-0.65 to -0.19] — A two-sided 95% CI of the estimated mean change from Baseline in hemoglobin was derived from the t-distribution
Statistical Analysis 2: Comparison: Peginesatide - Not on Dialysis; Test type: Superiority or Other; Mean change from baseline = 0.49, 95% CI 2-sided [0.26 to 0.71] — A two-sided 95% CI of the estimated mean change from Baseline in hemoglobin was derived from the t-distribution

2. Secondary Outcome: Percentage of Participants With Hemoglobin Within the Target Range of 10.0 to 12.0 g/dL During the Evaluation Period
Description: Mean hemoglobin was calculated from measurements taken during the Evaluation Period from Week 19 to Week 24. The target hemoglobin range was between 10.0 to 12.0 g/dL.
  The 95% confidence interval was calculated from the normal approximation with continuity correction.
Time Frame: Week 19 to Week 24
Population: Full Analysis Set where data was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginesatide - On Dialysis | Peginesatide - Not on Dialysis
Number analyzed (Participants) | 45 | 47
percentage of participants | 73.3 [59.3 to 87.4] | 68.1 [53.7 to 82.5]

3. Secondary Outcome: Percentage of Participants With a Change in Hemoglobin From Baseline to the Evaluation Period Within 1 g/dL
Description: Percentage of participants with a mean change in hemoglobin between Baseline (the mean of the 4 most recent hemoglobin values prior to enrollment and the hemoglobin on the day of enrollment) and the Evaluation Period (mean hemoglobin measured at Weeks 19 to 24) of less than or equal ± 1 g/dL.
  The 95% confidence interval was calculated from the normal approximation with continuity correction.
Time Frame: Baseline and Week 19 to Week 24.
Population: Full analysis set where data was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginesatide - On Dialysis | Peginesatide - Not on Dialysis
Number analyzed (Participants) | 45 | 47
percentage of participants | 80.0 [67.2 to 92.8] | 68.1 [53.7 to 82.5]

4. Secondary Outcome: Percentage of Participants With Red Blood Cell Transfusions
Description: The percentage of participants who received one or more red blood cell transfusions, including packed red blood cells and whole blood transfusions, during the Titration Period (Weeks 0 - 18) and Evaluation Period (Weeks 19 -24). 95% Confidence Intervals were calculated from the normal approximation with continuity correction.
Time Frame: Up to 24 weeks.
Population: Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginesatide - On Dialysis | Peginesatide - Not on Dialysis
Number analyzed (Participants) | 52 | 49
percentage of participants
  Entire study | 5.8 [0.0 to 13.1] | 2.0 [0.0 to 7.0]
  Titration Period | 5.8 [0.0 to 13.1] | 2.0 [0.0 to 7.0]
  Evaluation Period | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]

5. Secondary Outcome: Mean Hemoglobin During 4-week Intervals
Description: Hemoglobin was measured every 2 weeks during the Titration Period (Weeks 0-18) and weekly during the Evaluation Period (Weeks 19-24).
Time Frame: Up to 24 weeks.
Population: Full Analysis Set where data was available for each time interval (indicated by N).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Peginesatide - On Dialysis | Peginesatide - Not on Dialysis
Number analyzed (Participants) | 52 | 49
g/dL
  Week 1-4 [N=52, 49] | 11.54 (0.728) | 11.74 (0.863)
  Week 5-8 [N=49, 49] | 11.16 (0.876) | 11.94 (0.917)
  Week 9-12 [N=49, 47] | 10.99 (0.919) | 11.95 (0.837)
  Week 13-16 [N=47, 46] | 10.64 (0.975) | 11.95 (0.815)
  Week 17-20 [N=46, 47] | 10.78 (0.989) | 11.84 (0.747)
  Week 21-24 [N=44, 47] | 10.81 (0.827) | 11.58 (0.687)

6. Secondary Outcome: Percentage of Participants With Target Hemoglobin of 10.0 to 12.0 g/dL by 4-week Intervals.
Description: Percentage of participants with mean hemoglobin levels falling between the target level of 10.0 to 12.0 g/dL during 4-week study intervals. Hemoglobin was measured every 2 weeks during the Titration Period (Weeks 0-18) and weekly during the Evaluation Period (Weeks 19-24). 95% Confidence Intervals were calculated from the normal approximation with continuity correction.
Time Frame: Up to 24 weeks.
Population: Full analysis set where data was available for each time interval (indicated by N).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginesatide - On Dialysis | Peginesatide - Not on Dialysis
Number analyzed (Participants) | 52 | 49
percentage of participants
  Week 1-4 [N=52, 49] | 71.2 [57.9 to 84.4] | 69.4 [55.5 to 83.3]
  Week 5-8 [N= 49, 49] | 81.6 [69.8 to 93.5] | 51.0 [36.0 to 66.0]
  Week 9-12 [N= 49, 47] | 77.6 [64.8 to 90.3] | 44.7 [29.4 to 60.0]
  Week 13-16 [N= 47, 46] | 74.5 [60.9 to 88.0] | 52.2 [36.7 to 67.7]
  Week 17-20 [N=46, 47] | 69.6 [55.2 to 83.9] | 59.6 [44.5 to 74.7]
  Week 21-24 [N=44, 47] | 79.5 [66.5 to 92.6] | 63.8 [49.0 to 78.6]

7. Secondary Outcome: Percentage of Participants With Dose Adjustments During the Study
Description: The peginesatide dose was adjusted to maintain Hemoglobin values in the target range of 10 to 12 g/dL and ±1.5 g/dL from Baseline during the Titration Period (Weeks 0-18) and Evaluation Period (Weeks 19-24). A dose was classified as adjusted if it was not within 20% of the previous dose. A dose was classified as increased or decreased if it was >20% higher or >20% lower respectively, than the previous dose.
Time Frame: From Week 4 to Week 20
Population: Safety Analysis set, which included all patients who received at least 1 dose of study drug. N indicates the number of patients with study drug administered during the period after excluding the initial dose of study drug and excluding the first dose after a restart of study drug and is the denominator for percentage calculations.
Measure: Number; unit: percentage of participants
Groups:
- IV Peginesatide - On Dialysis: Participants on dialysis received 0.04 to 0.16 mg/kg Peginesatide intravenous (IV) injection once every 4 weeks for 24 weeks. Initial dose based on patient's previous total weekly darbepoetin alfa dose, and thereafter could be adjusted to maintain hemoglobin values in the target range of 10 to 12 g/dL and ±1.5 g/dL from Baseline.
- SC Peginesatide - On Dialysis: Participants on dialysis received 0.04 to 0.16 mg/kg Peginesatide subcutaneous (SC) injection, once every 4 weeks for 24 weeks. Initial dose based on patient's previous total weekly darbepoetin alfa dose, and thereafter could be adjusted to maintain hemoglobin values in the target range of 10 to 12 g/dL and ±1.5 g/dL from Baseline.
- Peginesatide - Not on Dialysis: Participants not on dialysis received 0.04 to 0.16 mg/kg Peginesatide subcutaneous injection, once every 4 weeks for 24 weeks. Initial dose based on patient's previous total weekly darbepoetin alfa dose, and thereafter could be adjusted to maintain hemoglobin values in the target range of 10 to 12 g/dL and ±1.5 g/dL from Baseline.
Arm/Group | IV Peginesatide - On Dialysis | SC Peginesatide - On Dialysis | Peginesatide - Not on Dialysis
Number analyzed (Participants) | 47 | 5 | 49
percentage of participants
  Any adjustment in Titration Period [N=44, 5, 49] | 81.8 | 80.0 | 81.6
  Any adjustment in Evaluation Period [N=38, 5, 44] | 31.6 | 60.0 | 43.2
  Any adjustment during entire study [N=44, 5, 49] | 90.9 | 80.0 | 87.8
  Dose increased in Titration Period [N=44, 5, 49] | 56.8 | 40.0 | 10.2
  Dose increased in Evaluation Period [N=38, 5, 44] | 21.1 | 40.0 | 2.3
  Dose increased during entire study [N=44, 5, 49] | 65.9 | 60.0 | 12.2
  Dose decreased in Titration Period [N=44, 5, 49] | 50.0 | 60.0 | 73.5
  Dose decreased in Evaluation Period [N=38, 5, 44] | 13.2 | 20.0 | 40.9
  Dose decreased during entire study [N=44, 5, 49] | 59.1 | 60.0 | 79.6

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that occurred on or after the day of the first dose of peginesatide injection through the Follow-up phone call, which occurred within 28 days after the last dose.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Peginesatide - On Dialysis | Peginesatide - Not on Dialysis
Serious Adverse Events (participants affected / at risk) | 16/52 | 6/49
Other Adverse Events (participants affected / at risk) | 31/52 | 28/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide - On Dialysis (N=52) | Peginesatide - Not on Dialysis (N=49)
Cardiac failure congestive (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Dermo-hypodermitis (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — This treatment-emergent death occured during titration period and is not related.
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 — This treatment-emergent death occured during titration period and is not related.
Renal failure acute (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic valve replacement (Surgical and medical procedures) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide - On Dialysis (N=52) | Peginesatide - Not on Dialysis (N=49)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 6
Nausea (Gastrointestinal disorders) | 6 | 3
Consitpation (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 6 | 0
Oedema Peripheral (General disorders) | 2 | 6
Astenia (General disorders) | 1 | 3
Chest Discomfort (General disorders) | 3 | 0
Injection Site Extravasation (General disorders) | 3 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 6
Sinusitis (Infections and infestations) | 0 | 3
Thrombosis in Device (Injury, poisoning and procedural complications) | 4 | 0
Vascular Graft Complication (Injury, poisoning and procedural complications) | 3 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 7 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 2 | 5
Headache (Nervous system disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypertension (Vascular disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.